CLINICAL TRIAL: NCT05847361
Title: Can bh4 Levels Predict Severity and Complications of Pre Eclampsia in Pregnant Women
Brief Title: BH4 Blood Levels Variations in Pre Eclamptic Women
Acronym: BH4P
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, associate professor, University Tunis El Manar
Other Study IDs: Tunis Elmanar university
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Pre Eclampsia; Eclampsia, Antepartum; HELLP Syndrome (HELLP), Unspecified Trimester; Acute Renal Failure; Abruptio Placentae; Complicating Pregnancy
Keywords: BH4; Pre eclampsia; pregnancy; cesarean section
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; HELLP Syndrome; Acute Kidney Injury; Abruptio Placentae; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P: (P) : Preclamptic women : pregnant women diagnosed with preclampsia
  Interventions: Diagnostic Test: BH4 blood level
- N: (N) : normotensive women : pregnant women without any criteria of preeclampsia
  Interventions: Diagnostic Test: BH4 blood level

INTERVENTIONS:
Diagnostic Test: BH4 blood level — from admission to END OF PREGNANCY, a blood sample is taken.

SUMMARY:
tetrahydrobiopterin (BH4) is degraded by several enzymes, including BH4 oxidase and peroxidases. Several factors can affect its synthesis and degradation. BH4 deficiency or depletion and genetic variations in the genes involved in BH4 metabolism have been associated with hypertension, suggesting that BH4 may play a role in the pathogenesis of hypertension.

The maternity center of Tunis ( CMNT ) is a level 3 maternity center, supporting over 12 000 births yearly, where the caesarean section's rate is very high, close to 45% of deliveries.

Early detection of these patients can help control maternal and neonatal safety outcomes. we can avoid complications such as severe preeclampsia, HELLP syndrom and eclampsia for the mother, and preterm delievery and fetal growth restriction for the new born.

in the literature, studies have reported a decrease in BH4 levels in pregnant women compared to non-pregnant women and others showed that its deficiency or depletion has been associated with hypertension. Moreover, tetrahydrobiopterin administration has been studied as a potential treatment for preeclampsia but the optimal dose has not yet been determined, and further studies are needed to determine the appropriate dose, timing, and duration of BH4 supplementation in this context.

Thus, BH4 blood levels as a mean of screening, could enrich our diagnostic arsenal. The purpose of our study is to compare BH4 levels between preeclamptic and normotensive women.

DETAILED DESCRIPTION:
The investigators will conduct a monocentric , prospective, observational study, including 300 pregnant women (150 normotensive and 150 preeclamptic).

The participants will be divided into 2 equal groups :

* Group P : Preclampsia
* Group N : Normotensive

After written and informed consent are obtained, a standard battery of blood tests including serum BH4 will be runned for the eligible patients at any moment from the admission to the end of the pregnancy.

Baseline data will be collected at enrollment, including demographic and medical history information, blood pressure, proteinuria, and blood samples for BH4 and other biomarker measurements. Follow-up data will be collected at delivery, including blood pressure, proteinuria, and fetal growth measurements, as well as maternal and neonatal outcomes;

After collecting all groups, blood samples will be analysed for BH4.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 18 YEARS
* informed consent
* Pregnant
* Term of pregnancy over than 24 weeks of gestation
* Having a normal pregnancy ( for the control group)
* Being diagnosed with preeclampsia or severe preeclampsia as defined in international guidelines (for the case group)

Non- inclusion Criteria:

* Women with known phenylketonuria
* Any history of ( treated or not) hypertension prior to the current pregnancy
* Any history of ( treated or not) diabetes or gestational diabetes during the current pregnancy
* Any history of renal failure or kidney injury) in the current pregnancy
* Women under long-term medications for arterial hypertension or before 24 week of the current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 parturients free from any exclusion criteria , devided equally into 2 groups :
  Group P : Preclamptic women : pregnant women in which the diagnosis of preclampsia have been sustaiend
  Group N : Normotensive women : pregnant women without any criteria of preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
the association between BH4 blood level (ng/mL) and severity of preeclampsia (biological and clinical criteria) | From date of first admission until the date of foetal extraction, starting from 20 weeks of pregnancy to it's end (Maximal time frame : 22 weeks)
  The primary outcome measure will be the association between BH4 levels and the severity of preeclampsia, including maternal and fetal complications Preeclampsia is defined by : Systolic blood pressure (SBP) higher than 140 mmHg or/and diastolic blood pressure (DBP)higher than 90 mmHg whith proteinuria higher than 0.3 g/24 h
  Its sevrity is defined by at least one of those criteria:
  * SBP > 160 mmHg and/or DBP >110 mmHg
  * proteinuria > 3g/24h
  * creatini level > 90 µmol/ l
  * oliguria < 500 ml /24 hours or < 25 ml/ h
  * thrombocytopenia < 100.000/mm3
  * Cytolysis > two times the normal value
  * neurosensory signs
  * chest pain , acute lung edema, dyspnea

SECONDARY OUTCOMES:
the association between BH4 blood level (ng/mL) and gestational hypertension. | From date of first admission until the date of foetal extraction, starting from 20 weeks of pregnancy to it's end (Maximal time frame : 22 weeks)
  Secondary outcome measures will include the associationtion between BH4 levels and gestational hypertension.
  gestational hypertension are defined by High Blood pressure SBP > 160 mmHg and/or DBP > 90 mmHg without proteinuria or any other preeclamptic criteria

OTHER OUTCOMES:
the association between BH4 blood level (ng/mL) and preterm delivery (before 37 weeks of pregnancy) | From date of first admission until the date of foetal extraction, starting from 20 weeks of pregnancy to it's end (Maximal time frame : 22 weeks)
  Secondary outcome measures will include the predectivity of preterm delivery with BH4 levels
the association between BH4 blood level (ng/mL) and fetal growth restriction. | From date of first admission until the date of foetal extraction, starting from 20 weeks of pregnancy to it's end (Maximal time frame : 22 weeks)
  Secondary outcome measures will include the association between BH4 levels and fetal growth restriction.
the association between BH4 blood level (ng/mL) and placenta abroptio | From date of first admission until the date of foetal extraction, starting from 20 weeks of pregnancy to it's end (Maximal time frame : 22 weeks)
  econdary outcome measures will include the association between BH4 levels and placenta abroptio
the association between BH4 blood level (ng/mL) and mortality | From date of first admission until the date of foetal extraction, starting from 20 weeks of pregnancy to it's end (Maximal time frame : 22 weeks)
  predectivity of maternal and foetal mortality by BH4 levels

CONTACTS AND LOCATIONS:
Overall Officials: Hayen Magherbi, pr, Study Chair — faculty of medecine of tunis
Locations (1):
- Tunis maternity and neonatology center, minisetry of public health, Tunis, Tunisia